CLINICAL TRIAL: NCT02597686
Title: A Pilot Study of a Brief Self-distancing and Perspective Broadening Training Package for Bipolar Disorder
Brief Title: The STAGE Study for Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Collaborators: Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UEastAnglia
Record Dates: First submitted 2015-10-23; First posted 2015-11-05 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2015-11

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SD-PB training (Experimental)
  Interventions: Behavioral: SD-PB training

INTERVENTIONS:
Behavioral: SD-PB training

SUMMARY:
When the investigators are caught up in emotions, it is by stepping back (or decentering) that the investigators are able to see the situation from another perspective. Individuals with emotional disorders, however, can have difficulties in being able to do this.

Research has shown that improving an individual's ability to step back from their emotions and take perspective is possible and can have beneficial effects on depressive symptomatology (Self Distancing and Perspective Broadening [SDPB] training). The SDPB training package involves two techniques: 1) stepping back from situations using mental imagery (building a mental picture of the situation and changing the distance to it) and, 2) reframing situations using perspective broadening reappraisals (giving new meanings to situations). The training package trains these SDPB techniques using an individual's memories and every day events. The fortnightly training comprises of two one to one sessions and daily homework for a week in between.The SDPB training package is aimed at improving an individual's ability to step back from, and put a new meaning to emotional events that take place in their lives.

The prospective pilot study aims to investigate whether the SDPB training package reduces symptomatology and improves these abilities in individuals who experience both depressive and manic episodes (Bipolar Disorder [BD]).

BD has a cumulative lifetime prevalence ranging from 1.52% across Europe and is treated with moderate success using Cognitive Behavioural therapy (CBT). However, 'moderate success' is considerably low compared to other mental health problems and CBT can be time time consuming, expensive, and cognitively demanding (requiring a high level of functioning of one or more cognitive functions). Accordingly, BD may be one of the emotional disorders in greatest need of novel and evidence based treatments.

ELIGIBILITY:
Inclusion criteria include:

- Individuals with a diagnosis of Bipolar Disorder whom are at the time of testing in a euthymic state (not in an episode of depression or mania).

Exclusion criteria include:

* Current substance dependence or abuse
* Current CBT treatment
* Individuals who are not fluent in English
* Organic brain injury
* Active psychotic and manic symptoms requiring hospitalisation
* Active suicidal risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The Quick Inventory of Depressive Symptomatology | 21 days
  A modified daily measure of depressive symptoms
The Altman Self Rating Mania Scale | 21 days
  A modified daily measure of mania symptoms

SECONDARY OUTCOMES:
The Experiences Questionnaire | over 5 weeks
  A measure of the ability to decenter
The Cognitive Emotion Regulation Questionnaire | over 5 weeks
  A measure of the ability to perspective-take

CONTACTS AND LOCATIONS:
Locations (1):
- University of East Anglia, Doctorate in Clinical Psychology, Norwich, United Kingdom